CLINICAL TRIAL: NCT01279941
Title: Safety & Health Improvement: Enhancing Law Enforcement Departments
Acronym: SHIELD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kerry Kuehl, Associate Professor of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: e6309
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Physical Activity; Nutrition; Health Promotion; Stress, Psychological; Cardiovascular Diseases; Cancer
MeSH Terms: conditions — Motor Activity; Stress, Psychological; Cardiovascular Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testing Only (No Intervention)
- Testing & Intervention (Experimental)
  Interventions: Behavioral: Behavioral: Team-based intervention

INTERVENTIONS:
Behavioral: Behavioral: Team-based intervention — The intervention involves a scripted peer-taught interactive curriculum, which is delivered as twelve, one-hour weekly sessions incorporated into a team's usual work time activities, with four follow-up booster sessions after twelve months.
  Arms: Testing & Intervention

SUMMARY:
Researchers from Oregon Health & Science University have developed a science-based, team-centered, scripted peer-taught program for fire fighters improving diet and exercise behavior while reducing injury rates and costs. Those investigators are partnering with local law enforcement agencies in Oregon and SW Washington to adapt, apply and assess this work-based program among a new high risk group to improve the health and safety of law enforcement officers (LEOs). Fire fighters' work structure is a natural fit for a team-centered format, and teammates' social support appeared to partially mediate the intervention's positive outcomes. Although conducive to team formation, LEOs' work lacks the established team structure of fire fighters. This proposal will apply the team-centered intervention to LEOs and in the process, learn more about teams as vehicles of health behavior change, and their relationship with outcomes and other potential mediating variables in a multilevel ecological analytic framework.

DETAILED DESCRIPTION:
Following a 3 month pilot study with four teams, we will enroll 14 precincts and 80 teams (approximately 470 participants) of LEO work groups for a prospective, clustered randomized 2-year assessment of the intervention (40 intervention and 40 testing-only, control-condition teams). Participants will be evaluated at baseline, 12, and 24. Primary study aims are; 1) Implement a randomized controlled efficacy trial of the SHIELD intervention, a peer-led, team-based occupational wellness program, and assess its behavioral and occupational outcomes, 2) Determine relations among variables in the chain from exposure of LEO subjects to specific intervention components to changes in mediating variables to behavior changes and occupational outcomes, and 3) Perform a cost analysis to determine the economic benefit of this LEO worksite health promotion program.

The intervention involves a scripted peer-taught interactive curriculum, which is delivered as twelve, one-hour weekly sessions incorporated into a team's usual work time activities, with four follow-up booster sessions after twelve months. The curriculum is designed to build understanding, healthy decision making skills and engender the social support of teammates; its content and scope reflects the core lifestyles activities used with fire fighters, along with adaptations for the needs of LEOs in domains of the team-building, family support and psychological health.

Participant assessments include established survey instruments, physiological measures and selected laboratory parameters of outcomes and potential mediating variables at the individual, interpersonal and organizational levels. Intervention delivery and fidelity will be assessed. Multilevel and latent growth modeling and mediation analyses will be used to assess outcomes and the relationships among variables. At proposal completion there will be an evidenced-based, exportable occupational safety and health program for LEOs. Its critical components will be defined, and its benefits clearly determined.

ELIGIBILITY:
Inclusion Criteria:

* member of a participating Law Enforcement Organization

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2010-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
BMI | January 2011-Dec 2014
Fruit and Vegetable Intake | January 2011-Dec 2014
Physical Activity | January 2011-Dec 2014
Stress | January 2011-Dec 2014
Sleep | January 2011-Dec 2014
Alcohol Use | January 2011-Dec 2014
Tobacco Use | January 2011-Dec 2014

SECONDARY OUTCOMES:
Blood Pressure | January 2011-Dec 2014
Percent Body Fat | January 2011-Dec 2014
Lipids and Lipoproteins | January 2011-Dec 2014
Glucose | January 2011-Dec 2014
Fasting Insulin | January 2011-Dec 2014
Cost-Effective Analysis | January 2011-Dec 2014

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Kuehl, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States